CLINICAL TRIAL: NCT01982162
Title: Protocol for the European Multi-Centre Study Understanding Severe Asthma Longitudinal Assessment of Children With Severe Asthma and Severe Pre-school Wheeze
Brief Title: Longitudinal Assessment of Children With Severe Asthma and Severe Pre-school Wheeze
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. P.J. Sterk, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 10/H0801/65
Record Dates: First submitted 2013-10-30; First posted 2013-11-13 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Asthma
Keywords: Sputum; Clinical cohorts; Smokers; Asthma; Biopsies; Severe asthma; Collaborative research; Phenotyping; Lipidomics; Transcriptomics; Proteomics; Paediatric cohort; Systems Biology
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort A: severe school aged asthma cohort
- Cohort B: mild to moderate school aged asthma cohort
- Cohort C: Severe pre school wheeze cohort
- Cohort D: Mild to moderate pre school wheeze cohort

SUMMARY:
Cross-sectional study to characterize cohorts of children with asthma and healthy controls in terms of clinical features, physiological measurements and non-invasive measurement of biomarkers and develop phenotype handprints for children with severe asthma

ELIGIBILITY:
Inclusion Criteria:

1. Parent / guardian must be able to give written informed consent prior to participation in the study, which includes ability to comply with the requirements and restrictions listed in the consent form. Informed consent must be obtained prior to undertaking any study procedures.
2. Assent should be obtained from all children in the study where appropriate.
3. Male or female subject aged between 1 - 17 years inclusive at screening.
4. The parent / guardian, or where appropriate the child must be able to read, comprehend, and write at a sufficient level to complete study related materials.
5. Subjects will be allowed to enrol in other studies while taking part on this study. However, Permission from the Scientific Board must be obtained to enrol or allow the continued participation of a subject enrolled in another study.

Exclusion Criteria:

1. As a result of medical interview, physical examination or screening investigation the physician responsible considers the child unfit for the study.
2. The subject has a history of drug or other allergy, which, in the opinion of the responsable physician, contra-indicates their participation.
3. Subject is female who is pregnant or lactating or up to 6 weeks post partum or 6 weeks cessation of breast feeding. If a woman is subsequently found to have been pregnant at the time of an assessment data from that assessment will not be included in the analyses
4. The child has participated within 3 months of the first dose in a study using a new molecular entity, or the first dose in any other study investigating drugs or having participated within three months in a study with invasive procedures. Any U-BIOPRED assessments should be deferred until 3 months after the first dose or invasive procedure. Permission from the Scientific Board must be obtained to enroll or allow the continued participation of a child enrolled in another study.
5. Those who, in the opinion of the investigator, have a risk of non-compliance with study procedures.
6. Prematurity ≤35 weeks gestation
7. The child had changed asthma medication within 4 weeks of the screening assessment(except those using the Symbicort maintenance and reliever therapy (SMART) regime)(assessment should be deferred)
8. History or current evidence of an upper or lower respiratory infection or symptoms (including common cold) within 2 weeks of baseline assessment (assessment should be deferred).
9. The child has had a severe exacerbation (requiring ER attendance or hospital admission and/or a course of high dose OCS for at least 3 days duration) within 4 weeks of the baseline assessment (assessment should be deferred).

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * Severe school aged asthma cohort: persistent symptoms or frequent severe exacerbations or persistent airflow limitation
  * Mild-moderate school aged asthma cohort: controlled or partially controlled asthma symtomps
  * Severe pre school wheeze cohort: persistent symptoms or frequent severe exacerbations
  * Mild-moderate pre school wheeze cohort: controlled symptoms or partially controlled
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbations | 3 years
Lung function decline over the course of the study | 3 years
Changes in asthma medication | 3 years
Daily symptoms and short acting beta agonist (SABA) usage | 3 years
Asthma control questionnaire (ACQ) at baseline and changes over the course of the study | 3 years
Upper airway symptoms as assessed by the sino-nasal outcomes test (SNOT) at baseline and changes over the course of the study | 3 years
Sleep and daytime drowsiness as assessed by the Epworth sleepiness scale at baseline and changes over the course of the study | 3 years
Measurement of pulmonary function including spirometry, plethysmography, bronchodilator reversibility and respiratory impedance by forced oscillation technique | 3 years
Radiological parameters such as computerized tomography (CT) scan, including assessment of lung structure | 3 years
Measurement of inflammatory cell counts in blood, sputum and bronchoalveolar lavage (BAL) | 3 years
Histopathology of bronchial biopsies in a sub group of subjects | 3 years
Transcriptomics, proteomics and metabolomics will be used on samples such as blood, urine and endobronchial biopsies | 3 years
Quality of life as assessed by the asthma quality of life questionnaire (AQLQ) | 3 years
Anxiety and depression as assessed by the hospital anxiety and depression scale (HADS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans Bisgaard, Dr., Principal Investigator — Copenhaguen Unversity Hospital, Copenhaguen, Denmark; Gunila Hedlin, Dr., Principal Investigator — Astrid Lindgren Children's Hospital, Stockholm, Sweeden; Philip Latzin, Dr., Principal Investigator — Department Respiratory medicine Pediatrics Insespital University of Bern, Bern, Switzerland; Peter Sterk, Dr., Principal Investigator — Academic Medical Centre University of Amsterdam, Amsterdam, The Netherlands; Andrew Bush, Dr., Principal Investigator — Imperial College of London, London, UK; Graham Roberts, Dr., Principal Investigator — Southampton General Hospital, Southampton, UK; Claire Murray, Dr., Principal Investigator — Wythenshawe Hospital, Manchester, UK

REFERENCES:
- [Derived] Daud T, Roberts S, Zounemat Kermani N, Richardson M, Heaney LG, Adcock IM, Amrani Y, Bradding P, Siddiqui S. The Role of WNT5a and TGF-beta1 in Airway Remodelling and Severe Asthma. Allergy. 2025 Apr;80(4):1025-1037. doi: 10.1111/all.16445. Epub 2025 Jan 3. PMID 39749571
- [Derived] Rossios C, Pavlidis S, Hoda U, Kuo CH, Wiegman C, Russell K, Sun K, Loza MJ, Baribaud F, Durham AL, Ojo O, Lutter R, Rowe A, Bansal A, Auffray C, Sousa A, Corfield J, Djukanovic R, Guo Y, Sterk PJ, Chung KF, Adcock IM; Unbiased Biomarkers for the Prediction of Respiratory Diseases Outcomes (U-BIOPRED) Consortia Project Team. Sputum transcriptomics reveal upregulation of IL-1 receptor family members in patients with severe asthma. J Allergy Clin Immunol. 2018 Feb;141(2):560-570. doi: 10.1016/j.jaci.2017.02.045. Epub 2017 May 18. PMID 28528200
- [Derived] Loza MJ, Djukanovic R, Chung KF, Horowitz D, Ma K, Branigan P, Barnathan ES, Susulic VS, Silkoff PE, Sterk PJ, Baribaud F; ADEPT (Airways Disease Endotyping for Personalized Therapeutics) and U-BIOPRED (Unbiased Biomarkers for the Prediction of Respiratory Disease Outcome Consortium) investigators. Validated and longitudinally stable asthma phenotypes based on cluster analysis of the ADEPT study. Respir Res. 2016 Dec 15;17(1):165. doi: 10.1186/s12931-016-0482-9. PMID 27978840
- [Derived] Bigler J, Boedigheimer M, Schofield JPR, Skipp PJ, Corfield J, Rowe A, Sousa AR, Timour M, Twehues L, Hu X, Roberts G, Welcher AA, Yu W, Lefaudeux D, Meulder B, Auffray C, Chung KF, Adcock IM, Sterk PJ, Djukanovic R; U-BIOPRED Study Group ||. A Severe Asthma Disease Signature from Gene Expression Profiling of Peripheral Blood from U-BIOPRED Cohorts. Am J Respir Crit Care Med. 2017 May 15;195(10):1311-1320. doi: 10.1164/rccm.201604-0866OC. PMID 27925796
- [Derived] Fleming L, Murray C, Bansal AT, Hashimoto S, Bisgaard H, Bush A, Frey U, Hedlin G, Singer F, van Aalderen WM, Vissing NH, Zolkipli Z, Selby A, Fowler S, Shaw D, Chung KF, Sousa AR, Wagers S, Corfield J, Pandis I, Rowe A, Formaggio E, Sterk PJ, Roberts G; U-BIOPRED Study Group. The burden of severe asthma in childhood and adolescence: results from the paediatric U-BIOPRED cohorts. Eur Respir J. 2015 Nov;46(5):1322-33. doi: 10.1183/13993003.00780-2015. Epub 2015 Sep 24. PMID 26405287
- [Derived] Shaw DE, Sousa AR, Fowler SJ, Fleming LJ, Roberts G, Corfield J, Pandis I, Bansal AT, Bel EH, Auffray C, Compton CH, Bisgaard H, Bucchioni E, Caruso M, Chanez P, Dahlen B, Dahlen SE, Dyson K, Frey U, Geiser T, Gerhardsson de Verdier M, Gibeon D, Guo YK, Hashimoto S, Hedlin G, Jeyasingham E, Hekking PP, Higenbottam T, Horvath I, Knox AJ, Krug N, Erpenbeck VJ, Larsson LX, Lazarinis N, Matthews JG, Middelveld R, Montuschi P, Musial J, Myles D, Pahus L, Sandstrom T, Seibold W, Singer F, Strandberg K, Vestbo J, Vissing N, von Garnier C, Adcock IM, Wagers S, Rowe A, Howarth P, Wagener AH, Djukanovic R, Sterk PJ, Chung KF; U-BIOPRED Study Group. Clinical and inflammatory characteristics of the European U-BIOPRED adult severe asthma cohort. Eur Respir J. 2015 Nov;46(5):1308-21. doi: 10.1183/13993003.00779-2015. Epub 2015 Sep 10. PMID 26357963